CLINICAL TRIAL: NCT04965389
Title: A Study to Assess the Absolute Oral Bioavailability of Milvexian Using a 14C-Microtracer and Oral Solution in Healthy Participants With Additional Food Effect Comparison of a Spray-Dried Dispersion Formulation of Milvexian in Capsules
Brief Title: A Study of Milvexian Using an IV Microtracer With Additional Formulation and Food Effect Comparison in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV010-062; 2021-000892-35 (EudraCT Number)
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers
Keywords: Bioavailability; BMS-986177; 14C-Microtracer; Milvexian
MeSH Terms: interventions — milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment Sequence 1 (Experimental)
  Interventions: Drug: BMS-986177 Oral Solution; Drug: [14C]BMS-986177 Solution for Infusion; Drug: BMS-986177 Spray-dried Dispersion Capsules
- Treatment Sequence 2 (Experimental)
  Interventions: Drug: BMS-986177 Oral Solution; Drug: [14C]BMS-986177 Solution for Infusion; Drug: BMS-986177 Spray-dried Dispersion Capsules
- Treatment Sequence 3 (Experimental)
  Interventions: Drug: BMS-986177 Oral Solution; Drug: [14C]BMS-986177 Solution for Infusion; Drug: BMS-986177 Spray-dried Dispersion Capsules
- Treatment Sequence 4 (Experimental)
  Interventions: Drug: BMS-986177 Oral Solution; Drug: [14C]BMS-986177 Solution for Infusion; Drug: BMS-986177 Spray-dried Dispersion Capsules

INTERVENTIONS:
Drug: BMS-986177 Oral Solution — Specified dose on specified days
  Other Names: Milvexian, JNJ-70033093
Drug: [14C]BMS-986177 Solution for Infusion — Specified dose on specified days
Drug: BMS-986177 Spray-dried Dispersion Capsules — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the absolute oral bioavailability (amount of drug entering the bloodstream) of spray-dried dispersion (SDD) milvexian capsules in the fed and fasted states, and to bridge the exposures seen using only the oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body mass index (BMI) of 18.0 to 32.0 kg/m², inclusive. BMI = weight (kg)/ (height [m])²

Exclusion Criteria:

* History of gastrointestinal (GI) disease, upper or lower GI bleeding within 6 months, intracranial bleeding, tumor, aneurysms
* History or evidence of abnormal bleeding or coagulation disorder and/or evidence of coagulopathy, prolonged or unexplained clinically significant bleeding, or frequent unexplained bruising or thrombus formation, or a history of spontaneous bleeding, such as epistaxis, or family history of coagulopathies
* Any acute or chronic medical illness considered clinically significant by the investigator
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory, neurological or psychiatric disorder, as judged by the investigator

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Nottingham, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence 1: ABCED: On Day 1 of Treatment Period 1 all participants will receive the (A) milvexian oral solution in the fasted state, followed 1 hour later by the intravenous (IV) [14C]milvexian microdose infused over 15 minutes. On Day 1 for Treatment Periods 2 to 5, participants will receive (B) milvexian SDD high dose capsules in the fasted state, (C) milvexian SDD low dose capsules in the fed state, (E) milvexian SDD high dose capsules in the fed state, and (D) milvexian SDD low dose capsules in the fasted state with a minimum of 72 hour washout in between each treatment period.
- Treatment Sequence 2: ACDBE: On Day 1 of Treatment Period 1 all participants will receive the (A) milvexian oral solution in the fasted state, followed 1 hour later by the intravenous (IV) [14C]milvexian microdose infused over 15 minutes. On Day 1 for Treatment Periods 2 to 5, participants will receive (C) milvexian SDD low dose capsules in the fed state, (D) milvexian SDD low dose capsules in the fasted state, (B) milvexian SDD high dose capsules in the fasted state, and (E) milvexian SDD high dose capsules in the fed state with a minimum of 72 hour washout in between each treatment period.
- Treatment Sequence 3: ADECB: On Day 1 of Treatment Period 1 all participants will receive the (A) milvexian oral solution in the fasted state, followed 1 hour later by the intravenous (IV) [14C]milvexian microdose infused over 15 minutes. On Day 1 for Treatment Periods 2 to 5, participants will receive (D) milvexian SDD low dose capsules in the fasted state, (E) milvexian SDD high dose capsules in the fed state, (C) milvexian SDD low dose capsules in the fed state, (B) milvexian SDD high dose capsules in the fasted state with a minimum of 72 hour washout in between each treatment period.
- Treatment Sequence 4: AEBDC: On Day 1 of Treatment Period 1 all participants will receive the (A) milvexian oral solution in the fasted state, followed 1 hour later by the intravenous (IV) [14C]milvexian microdose infused over 15 minutes. On Day 1 for Treatment Periods 2 to 5, participants will receive (E) milvexian SDD high dose capsules in the fed state, (B) milvexian SDD high dose capsules in the fasted state, (D) milvexian SDD low dose capsules in the fasted state, (C) milvexian SDD low dose capsules in the fed state with a minimum of 72 hour washout in between each treatment period.
Period: Overall Study
Arm/Group | Treatment Sequence 1: ABCED | Treatment Sequence 2: ACDBE | Treatment Sequence 3: ADECB | Treatment Sequence 4: AEBDC
Started (Started = Randomized) | 4 | 5 | 4 | 4
Participants Completed Treatment Period 1 | 4 (Treatment A=Oral solution with IV microdose) | 5 (Treatment A=Oral solution with IV microdose) | 4 (Treatment A=Oral solution with IV microdose) | 4 (Treatment A=Oral solution with IV microdose)
Participants Completed Treatment Period 2 | 4 (Treatment B=high dose milvexian SDD fasted) | 4 (Treatment C=low dose milvexian SDD fed) | 4 (Treatment D=low dose milvexian SDD fasted) | 4 (Treatment E=high dose milvexian SDD fed)
Participants Completed Treatment Period 3 | 3 (Treatment C=low dose milvexian SDD fed) | 4 (Treatment D=low dose milvexian SDD fasted) | 4 (Treatment E=high dose milvexian SDD fed) | 4 (Treatment B=high dose milvexian SDD fasted)
Participants Completed Treatment Period 4 | 3 (Treatment E=high dose milvexian SDD fed) | 3 (Treatment B=high dose milvexian SDD fasted) | 4 (Treatment C=low dose milvexian SDD fed) | 4 (Treatment D=low dose milvexian SDD fasted)
Participants Completed Treatment Period 5 | 3 (Treatment D=low dose milvexian SDD fasted) | 3 (Treatment E=high dose milvexian SDD fed) | 4 (Treatment B=high dose milvexian SDD fasted) | 4 (Treatment C=low dose milvexian SDD fed)
Completed (Completed=completed the study) | 3 | 3 | 4 | 4
Not Completed | 1 | 2 | 0 | 0
Not completed — Other reasons | 1 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 1 | 0 | 0
Not completed — Poor/Non-compliance | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: ABCED | Treatment Sequence 2: ACDBE | Treatment Sequence 3: ADECB | Treatment Sequence 4: AEBDC | Total
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.0 (14.5) | 45.4 (10.1) | 45.8 (15.0) | 37.3 (16.2) | 42.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 0 | 4
  Male | 3 | 4 | 2 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 4 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 2
  White | 2 | 4 | 4 | 4 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Absolute Bioavailability (F)
Description: Absolute bioavailability is defined as the amount of drug from a formulation that reaches the systemic circulation relative to an intravenous (IV) dose. Treatment A (milvexian oral solution with IV microdose) was assessed versus each treatment phase of milvexian administered as: a oral solution (fasted), high dose SDD (Spray-Dried Dispersion) capsule (fed and fasted) and low dose SDD capsule (fed and fasted).
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: Evaluable PK population-all participants who received at least one dose of study drug and had any available concentration-time data with adequate PK profiles for accurate estimation of PK parameters
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage of drug
Groups:
- Treatment A: Oral Solution With IV: Milvexian oral solution with IV microdose
- Treatment B: High Dose SDD Fasted: High dose milvexian SDD (spray-dried dispersion) was administered to a fasted population
- Treatment C: Low Dose SDD Fed: Low dose milvexian SDD (spray-dried dispersion) fed
- Treatment D: Low Dose SDD Fasted: Low dose milvexian SDD (spray-dried dispersion) fasted
- Treatment E: High Dose SDD Fed: High dose milvexian SDD (spray-dried dispersion) fed
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 14
Percentage of drug | 105 [103 to 109] | 54.2 [48.9 to 63.7] | 44.3 [39.6 to 53.0] | 58.2 [52.8 to 70.7] | 75.6 [71.1 to 81.8]

2. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: The number of participants experiencing AEs following single oral and IV administration. AEs are defined as any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 11 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Treatment B: High Dose SDD Fasted: High dose milvexian SDD (spray-dried dispersion) fasted
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 17 | 15 | 15 | 15 | 14
Participants
  Total participants with an adverse event | 8 | 2 | 2 | 0 | 2
  Adverse events leading to discontinuation | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAE)
Description: The number of participants experiencing SAEs following single oral and IV administration. SAEs are defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or causes prolongation of existing hospitalization.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 11 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 17 | 15 | 15 | 15 | 14
Participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Experiencing Abnormal Vital Sign Measurements
Description: Occurrence of abnormalities in vital sign measurements exceeding pre-defined thresholds following single oral and IV administration. The pre-defined thresholds include:
  Heart Rate(bpm) Value > 100 and change from baseline > 30, or Value < 55 and change from baseline < -15 Systolic Blood Pressure(mmHg) Value > 140 and change from baseline > 20, or Value < 90 and change from baseline < -20 Diastolic Blood Pressure(mmHg) Value > 90 and change from baseline > 10, or Value < 55 and change from baseline < -10 Respiratory Rate(breaths/min) Value > 16 or change from baseline > 10 Temperature (°C) Value > 38.3°C or change from baseline > 1.6°C
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 17 | 15 | 15 | 15 | 14
Participants
  Heart Rate (bpm) Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0 | 0
  Heart Rate (bpm) Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure (mmHg) Value > 140 and change from baseline > 20 | 0 | 0 | 1 | 0 | 0
  Systolic Blood Pressure (mmHg) Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0 | 1
  Diastolic Blood Pressure (mmHg) Value > 90 and change from baseline > 10 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) Value < 55 and change from baseline < -10 | 0 | 2 | 1 | 0 | 1
  Respiratory Rate (breaths/min) Value > 16 or change from baseline > 10 | 13 | 10 | 10 | 9 | 7
  Temperature (°C)Value > 38.3°C or change from baseline > 1.6°C | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs)
Description: The number of participants with abnormal findings on ECGs following single oral and IV administration. Participants with ECG intervals outside of a pre-specified range and investigator identified ECG abnormalities will be listed. The following criteria will be used to determine ECG results that are outside of a pre-specified range:
  PR (msec)-Value > 200; QRS (msec)-Value > 120; QT (msec)-Value > 500 or change from baseline > 30; QTcF (msec)-Value > 450 or change from baseline > 30
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 17 | 15 | 15 | 15 | 14
Participants | 2 | 2 | 1 | 0 | 1

6. Secondary Outcome: Number of Participants With Abnormal Physical Examinations
Description: The number of participants with abnormal findings on physical examinations following single oral and IV administration.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 17 | 15 | 15 | 15 | 14
Participants | 0 | 2 | 0 | 1 | 0

7. Secondary Outcome: Number of Participants With Clinical Laboratory Test Abnormalities
Description: Number of participants with abnormalities in clinical lab test measurements exceeding pre-defined thresholds following single oral and IV administration. The pre-defined thresholds include:
  Alanine transaminase > 3 × upper limit of normal (ULN) Aspartate transaminase > 3 × ULN Alkaline phosphatase > 1.5 × ULN Total bilirubin > 2 × ULN
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 17 | 15 | 15 | 15 | 14
Participants
  Alanine transaminase > 3 × upper limit of normal (ULN) | 0 | 0 | 0 | 0 | 0
  Aspartate transaminase > 3 × ULN | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase > 1.5 × ULN | 0 | 0 | 0 | 0 | 0
  Total bilirubin > 2 × ULN | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax is defined as the maximum observed plasma concentration following single administration in the fed and fasted states to healthy participants.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 14
ng/mL | 2929 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25.3 | 1200 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 31.0 | 130 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40.6 | 185 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 34.7 | 1696 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24.5

9. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax)
Description: Tmax is defined as the time of maximum observed plasma concentration in the fed and fasted states to healthy participants.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 14
Hours | 1.27 [0.500 to 4.00] | 4.00 [1.50 to 5.00] | 4.00 [1.00 to 6.00] | 4.00 [1.25 to 6.00] | 5.00 [4.00 to 10.0]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration [AUC(0-T)]
Description: AUC(0-T) is defined as the area under the plasma concentration-time curve from time zero to time of last quantifiable concentration following single administration in the fed and fasted states to healthy participants.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 14
ng.h/mL | 30844 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24.2 | 15855 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 33.4 | 1603 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 51.2 | 2183 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 60.6 | 21972 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25.1

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity [AUC(INF)]
Description: AUC(INF) is defined as area under the concentration-time curve from time zero extrapolated to infinity following single administration in the fed and fasted states to healthy participants
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 14
ng.h/mL | 31435 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25.3 | 16464 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 35.6 | 1569 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40.0 | 2061 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 32.6 | 22496 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28.6

12. Secondary Outcome: Apparent Clearance of Drug After Extravascular Administration (CLT/F)
Description: CLT/F is defined as the apparent clearance of drug after extravascular administration.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 14
Liters/hour | 6.36 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25.3 | 12.1 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 36.9 | 15.9 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 39.1 | 12.1 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 44.0 | 8.89 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 26.1

13. Secondary Outcome: Renal Clearance (CLR)
Description: CLR is defined as the volume of plasma completely cleared of a substance by the kidneys per unit of time, in this case by hour.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 14
Liters/hour | 1.63 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 31.3 | 1.68 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 31.6 | 1.91 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 29.0 | 1.84 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 27.4 | 1.70 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 30.3

14. Secondary Outcome: Apparent Volume of Distribution at Terminal Phase After Extravascular Administration (Vz/F)
Description: Vz/F is defined as the apparent volume of distribution at terminal phase after extravascular administration.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 14
Liters | 121 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25.8 | 243 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 37.2 | 344 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40.9 | 245 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 45.1 | 159 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 15.3

15. Secondary Outcome: Total Amount of Unchanged Drug Excreted Into the Urine (Ae)
Description: Ae is defined as the total amount of unchanged drug excreted into the urine following single administration in the fed and fasted states to healthy participants
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 14
mg | 50.2 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21.7 | 26.7 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28.0 | 3.06 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 43.7 | 4.01 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 42.8 | 37.3 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 20.6

16. Secondary Outcome: Total Percent Urinary Recovery (%UR)
Description: %UR is defined as a percent or absolute amount of dose that is recovered in the urine as the unchanged drug.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of milvexian recovered
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 14
Percentage of milvexian recovered | 25.1 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21.7 | 13.3 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28.0 | 12.2 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 43.7 | 16.0 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 42.8 | 18.6 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 20.6

17. Secondary Outcome: Half-life (T-HALF)
Description: T-HALF is defined as the time required for half the quantity of a drug to be metabolized or eliminated by normal biological processes.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 14
Hours | 13.3 (2.02) | 14.3 (4.08) | 15.8 (6.13) | 14.5 (4.10) | 12.8 (3.65)

18. Secondary Outcome: Mean Residence Time (MRT) Following an IV Dose in Treatment A
Description: Mean residence time (MRT) represents the average time the drug stays in the body and is evaluated for the IV dose of Treatment A only.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of Treatment A with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Oral Solution With IV
Number analyzed (Participants) | 16
Hours | 14.8 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21.8

19. Secondary Outcome: Volume of Distribution at Steady State (Vss) Following an IV Dose in Treatment A
Description: Characterize the IV dose of Treatment A by Vss, which is defined as the apparent volume of distribution at steady state
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of Treatment A with evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Treatment A: Oral Solution With IV
Number analyzed (Participants) | 16
Liters | 99.1 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 15.9

20. Secondary Outcome: Relative Bioavailability (Frel) Based on Ratios of Cmax
Description: Point estimates and 90% CI for the ratio of geometric means for Cmax will be constructed for the comparison of each milvexian capsule treatment (Treatments B, C, D, and E) separately versus the oral solution (Treatment A). No data is reported for Treatment A because it is the comparison treatment.
  Relative bioavailability is defined as the amount of drug from a formulation that reaches the systemic circulation relative to a different formulation (non-IV) such as an oral solution. Cmax is defined as the maximum observed plasma concentration.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 14
ng/mL | NA [NA to NA] — Data is not provided for Treatment A because it is the comparator for the other treatments and therefore could not be compared to itself. | 0.403 [0.354 to 0.459] | 0.358 [0.307 to 0.418] | 0.510 [0.427 to 0.610] | 0.574 [0.524 to 0.629]

21. Secondary Outcome: Relative Bioavailability (Frel) Based on Ratios of AUC(0-T) and AUC(INF)
Description: Point estimates and 90% CI for the ratio of geometric means for AUC(0-T) and AUC(INF) will be constructed for the comparison of each milvexian capsule treatment (Treatments B, C, D, and E) separately versus the oral solution (Treatment A). No data is reported for Treatment A because it is the comparison treatment.
  Relative bioavailability is defined as the amount of drug from a formulation that reaches the systemic circulation relative to a different formulation (non-IV) such as an oral solution. AUC(0-T) is defined as the area under the plasma concentration-time curve from time zero to time of last quantifiable concentration. AUC(INF) is defined as area under the concentration-time curve from time zero extrapolated to infinity.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of study drug with evaluable concentration-time data
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 14
ng.h/mL
  AUC(0-T) | NA [NA to NA] — Data is not provided for Treatment A because it is the comparator for the other treatments and therefore could not be compared to itself. | 0.513 [0.446 to 0.591] | 0.425 [0.367 to 0.492] | 0.570 [0.466 to 0.697] | 0.716 [0.661 to 0.775]
  AUC(INF) | NA [NA to NA] — Data is not provided for Treatment A because it is the comparator for the other treatments and therefore could not be compared to itself. | 0.522 [0.455 to 0.600] | 0.436 [0.375 to 0.507] | 0.543 [0.453 to 0.651] | 0.720 [0.664 to 0.780]

22. Secondary Outcome: Food Effect Based on Ratios of Cmax Following an SDD Capsule Dose in Treatment B, C, D, and E
Description: Food effect analysis of the high and low dose SDD capsules based on ratios of Cmax. The food effect analysis will be run separately for each dose level. For the low dose level, low dose milvexian SDD fed (Treatment C) is the test treatment and low dose milvexian SDD fasted (Treatment D) is the reference treatment. For the high dose dose level, high dose milvexian SDD fed (Treatment E) is the test treatment and high dose milvexian SDD fasted (Treatment B) is the reference treatment.
  Cmax is defined as the maximum observed plasma concentration.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of Treatment B, C, D, or E with evaluable concentration-time data
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 15 | 15 | 14 | 14
ng/mL | 1197 [1039 to 1378] | 128 [105 to 156] | 185 [153 to 223] | 1709 [1521 to 1920]

23. Secondary Outcome: Food Effect Based on Ratios of AUC(0-T) and AUC(INF) Following an SDD Capsule Dose in Treatment B, C, D, and E
Description: Food effect with low and high dose SDD capsules based on ratios of AUC(0-T) and AUC(INF). The food effect analysis will be run separately for each dose level. For the low dose level, low dose milvexian SDD fed (Treatment C) is the test treatment and low dose milvexian SDD fasted (Treatment D) is the reference treatment. For the high dose level, high dose milvexian SDD fed (Treatment E) is the test treatment and high dose milvexian SDD fasted (Treatment B) is the reference treatment.
  AUC(0-T) is defined as the area under the plasma concentration-time curve from time zero to time of last quantifiable concentration.
  AUC(INF) is defined as area under the concentration-time curve from time zero extrapolated to infinity.
Time Frame: Day 1 of Treatment Periods 1-5 (up to approximately 7 weeks)
Population: All participants who received at least one dose of Treatment B, C, D, or E with evaluable concentration-time data
Measure: Geometric Mean (90% Confidence Interval); unit: ng.h/mL
Arm/Group | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
Number analyzed (Participants) | 15 | 15 | 14 | 14
ng.h/mL
  AUC(0-T) | 15871 [13678 to 18415] | 1592 [1287 to 1969] | 2170 [1763 to 2670] | 22171 [19578 to 25108]
  AUC(INF) | 16480 [14067 to 19307] | 1545 [1291 to 1848] | 2069 [1749 to 2447] | 22774 [19892 to 26073]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to study completion (up to approximately 11 weeks). Serious Adverse events and other adverse events were assessed from date of first dose to 30 days following date of last dose (up to approximately 11 weeks).
Arm/Group | Treatment A: Oral Solution With IV | Treatment B: High Dose SDD Fasted | Treatment C: Low Dose SDD Fed | Treatment D: Low Dose SDD Fasted | Treatment E: High Dose SDD Fed
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15 | 0/15 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/15 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 8/17 | 2/15 | 2/15 | 0/15 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Oral Solution With IV (N=17) | Treatment B: High Dose SDD Fasted (N=15) | Treatment C: Low Dose SDD Fed (N=15) | Treatment D: Low Dose SDD Fasted (N=15) | Treatment E: High Dose SDD Fed (N=14)
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT04965389/Prot_SAP_000.pdf